CLINICAL TRIAL: NCT04227821
Title: Hemodynamic Optimalization in Pediatric Critically Ill Patients: Prospective Observational Trial
Brief Title: Hemodynamic Optimalization in Pediatric Patients
Acronym: HOPED
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, Clinical Professor, Brno University Hospital
Other Study IDs: KDAR FN Brno 2020/2
Record Dates: First submitted 2020-01-08; First posted 2020-01-14 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Hemodynamic Instability
Keywords: Hemodynamic instability; vasopressor therapy; Pediatric patient; Norepinephrine; Epinephrine; Dobutamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemodynamically instable pediatric patients: Pediatric patients admitted to the pediatric intensive care unit with the need of vasopressor and/or inotrope therapy due to hemodynamic instability
  Interventions: Other: Vasopressor and/inotrope therapy

INTERVENTIONS:
Other: Vasopressor and/inotrope therapy — In pediatric patients admitted to the pediatric intensive care, with the persistent hemodynamic instability after fluid resuscitation, the vasopressor and/or inotrope therapy will be initiated
  Other Names: Hemodynamic optimalization

SUMMARY:
Hemodynamic unstability, defined by macrocirculation and/or microcirculation dysfunction or alteration is common in critically ill pediatric patients. The initial treatment of hemodynamically unstable patient is the fluid resuscitation (fluid challenge therapy). However, the stabilization of hemodynamics only with fluid resuscitation can be achieved in less than 50% pediatric patients. In case of persistent hypotension (defined as mean arterial pressure below 65 mmHg, or by the formula - 55 + 1,5 x age in years), or in case of persistent lactate levels and base deficit elevation is the catecholamine therapy method of choice in case of sufficiently restored intravascular volume. In adult patients, the drug of choice (the first line therapy of persistent hypotension) is considered norepinephrine (based on evidence-based data). The norepinephrine is administered intravenously in form of continuous infusion, with the dose adjusted to the target level of mean arterial pressure (MAP). It should be preferably administered through the central venous catheter to minimize the complications associated with the damage of the peripheral vein wall damage in case of administered into the peripheral vein. Due to lack of evidence-based data (EBM) for pediatric population, there is still significant heterogenity of clinical practice and dobutamin, dopamine, norepinephrine and epinephrine are being used for hemodynamically unstable pediatric patient.

DETAILED DESCRIPTION:
After Ethics committee approval, pediatric patients admitted to the Departement of pediatric anesthesiology and intensive care with the need of vasopressor and/or inotrope therapy in the selected study period will be included. The primary aim of the trial is the describe the therapy effect on the vital signs (heart rate, blood pressure), level of lactate and base deficit in 1,3,6,12,24,48 and every other 24th hours. The secondary aim of the trial is the incidence of complications: arrythmias, hypertension, defects of peripheral perfusion, mortality, renal failure, the PELOD-2 and pSOFA score at admission and every next 24 hours. The cumulative overall dose and the cumulative 24 hours dose of vasopressors/inotropes will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients in selected age interval
* admitted to the pediatric intensive care unit
* hemodynamic instability with the need for vasopressor and/or inotrope therapy

Exclusion Criteria:

* patients with no hemodynamic instability
* patients with achieved hemodynamic stability after fluid resuscitation

Ages: 29 Days to 19 Years | Sex: All
Age Groups: Child, Adult
Study Population: Critically ill pediatric patients admitted to the pediatric intensive care unit with persitent hemodynamic instability despite adequate volume resuscitation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Vasopressor and/or inotrope therapy effect on blood pressure | From date of ICU admission until the date of weaning from vasopressor and/or inotrope therapy, assessed up to 1 month
  Blood pressure will be measured during ICU stay
Vasopressor and/or inotrope therapy effect on levels of lactate | From date of ICU admission until the date of weaning from vasopressor and/or inotrope therapy, assessed up to 1 month
  blood levels of lactate will be measured during ICU stay
Vasopressor and/or inotrope therapy effect on blood levels of base deficit | From date of ICU admission until the date of weaning from vasopressor and/or inotrope therapy, assessed up to 1 month
  blood levels of base deficit will be measured during ICU stay
Vasopressor and/or inotrope therapy effect on heart rate | From date of ICU admission until the date of weaning from vasopressor and/or inotrope therapy, assessed up to 1 month
  Heart rate will be measured during ICU stay

SECONDARY OUTCOMES:
Incidence of associated complications | From date of ICU admission until the date of weaning from vasopressor and/or inotrope therapy, assessed up to 1 month
  The incidence of arrythmias, hypertension, defects of peripheral perfusion, renal failure will be measured during the therapy
Change in Pediatric Logistic Organ Dysfunction-2 (PELOD-2 score) | From date of ICU admission until the date of weaning from vasopressor and/or inotrope therapy, assessed up to 1 month
  The Pediatric Logistic Organ Dysfunction-2 (PELOD-2) score will be measured every day from ICU admission until ICU discharge
Change in The Pediatric Sequential Organ Failure Assessment (pSOFA) | From date of ICU admission until the date of weaning from vasopressor and/or inotrope therapy, assessed up to 1 month
  The Pediatric Sequential Organ Failure Assessment (pSOFA) score will be measured every day every day from ICU admission until ICU discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Brno University Hospital, Brno, South Moravian, Czechia

IPD SHARING:
Plan to Share IPD: Undecided